CLINICAL TRIAL: NCT01989572
Title: A Randomized, Placebo-Controlled Phase III Trial of Yeast Derived GM-CSF Versus Peptide Vaccination Versus GM-CSF Plus Peptide Vaccination Versus Placebo in Patients With "No Evidence of Disease" After Complete Surgical Resection of "Locally Advanced" and/or Stage IV Melanoma
Brief Title: Sargramostim, Vaccine Therapy, or Sargramostim and Vaccine Therapy in Preventing Disease Recurrence in Patients With Melanoma That Has Been Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2013-02101; NCI-2013-02101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB 500101; U10CA021115 (NIH); ECOG-4697; CDR0000067568; SWOG-E4697; 9546; E4697 (Other: Eastern Cooperative Oncology Group); E4697 (Other: CTEP); NCT00005034 (obsolete NCT alias)
Record Dates: First submitted 2013-11-18; First posted 2013-11-21 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Iris Melanoma; Medium/Large Size Posterior Uveal Melanoma; Mucosal Melanoma; Ocular Melanoma With Extraocular Extension; Recurrent Melanoma; Recurrent Uveal Melanoma; Small Size Posterior Uveal Melanoma; Stage IIA Cutaneous Melanoma AJCC v6 and v7; Stage IIA Uveal Melanoma AJCC v7; Stage IIB Cutaneous Melanoma AJCC v6 and v7; Stage IIB Uveal Melanoma AJCC v7; Stage IIC Cutaneous Melanoma AJCC v6 and v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIA Uveal Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIB Uveal Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IIIC Uveal Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Arm I (sargramostim, peptide vaccine) (Experimental): Patients receive sargramostim SC on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Sargramostim; Biological: Tyrosinase Peptide
- Arm II (sargramostim placebo, peptide vaccine) (Experimental): Patients receive sargramostim placebo SC on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Biological: Tyrosinase Peptide
- Arm III (sargramostim, peptide placebo) (Experimental): Patients receive sargramostim SC on days 1-14 and peptide placebo mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Biological: Sargramostim
- Arm IV (placebo, peptide placebo) (Placebo Comparator): Patients receive placebo SC on days 1-14 and peptide placebo on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo
- Arm V (sargramostim) (Experimental): Patients receive sargramostim SC on days 1-14.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Sargramostim
- Arm VI (sargramostim placebo) (Placebo Comparator): Patients receive sargramostim placebo SC on days 1-14.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given GM-CSF placebo SC
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (sargramostim placebo, peptide vaccine); Arm IV (placebo, peptide placebo); Arm VI (sargramostim placebo)
Other: Placebo — Given peptide placebo SC
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm III (sargramostim, peptide placebo); Arm IV (placebo, peptide placebo)
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
  Arms: Arm I (sargramostim, peptide vaccine); Arm III (sargramostim, peptide placebo); Arm V (sargramostim)
Biological: Tyrosinase Peptide — Given SC
  Other Names: Tyrosinase Peptides
  Arms: Arm I (sargramostim, peptide vaccine); Arm II (sargramostim placebo, peptide vaccine)

SUMMARY:
This randomized phase III trial studies sargramostim or vaccine therapy alone to see how well they work compared to sargramostim and vaccine therapy together in preventing disease recurrence in patients with melanoma that has been removed by surgery. Sargramostim may stimulate the immune system in different ways and stop tumor cells from growing. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. It is not yet known whether yeast derived sargramostim and vaccine therapy are more effective alone or together in preventing recurrence of melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival and disease-free survival of patients with completely resected stage IV melanoma or stage III melanoma with gross extranodal extension, satellites, and/or intransit lesions, treated with granulocyte macrophage colony-stimulating factor (GM-CSF) (sargramostim) vs. no GM-CSF, or other high risk patients listed in the eligibility section.

SECONDARY OBJECTIVES:

I. To compare, using a 2 x 2 factorial design, overall survival and disease-free survival of human leukocyte antigen (HLA)-A2 positive patients treated with peptide vaccination vs. no peptide vaccination.

II. The following descriptive evaluations of survival and disease-free survival are planned for the HLA-A2 positive patients: (1) GM-CSF plus peptide vaccination vs. peptide vaccination alone; (2) GM-CSF plus peptide vaccination vs. GM-CSF alone; (3) GM-CSF plus peptide vaccination vs. placebo.

III. Survival and disease-free survival of HLA-A2 positive patients not receiving peptide vaccination will be compared to that of HLA-A2 negative patients not receiving peptide vaccination.

IV. To determine the influence of GM-CSF on circulating dendritic cell numbers and subpopulations in peripheral blood of patients receiving and not receiving GM-CSF.

V. To determine, in HLA-A2 positive patients, whether immunization with peptides with or without GM-CSF elicits a measurable T-cell response as assessed by enzyme-linked immunosorbent spot (ELISPOT) and the major histocompatibility complex (MHC) tetramer assay, and to determine the functionality of these cells by intracellular cytokine staining.

OUTLINE: HLA-A2 positive patients are randomized to 1 of 4 treatment regimens (Arms I-IV). HLA-A2 negative patients are randomized to 1 of 2 treatment arms (Arms V-VI).

ARM I: Patients receive sargramostim subcutaneously (SC) on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).

ARM II: Patients receive sargramostim placebo SC on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).

ARM III: Patients receive sargramostim SC on days 1-14 and peptide placebo mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).

ARM IV: Patients receive sargramostim placebo SC on days 1-14 and peptide placebo mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).

ARM V: Patients receive sargramostim SC on days 1-14.

ARM VI: Patients receive sargramostim placebo SC on days 1-14.

In all arms, treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

In the event of recurrence, patients who undergo complete resection of the recurrence may continue treatment for 6 courses or until completion of 1 year of therapy (whichever is longer). For patients with recurrence that is not surgically resectable or experiencing second recurrence, treatment will be discontinued.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have HLA-A2 status known prior to randomization; typing may be obtained through a local laboratory facility or through a reference lab utilized by the initiating institution; if typing is not available through these means, it may be obtained from the University of Pittsburgh
* All patients must have disease completely resected with one of the following in order to be eligible:

  * Completely resected disease
  * Any locoregional recurrence after prior adjuvant interferon or failure on S008
  * Any local recurrence of disease after adequate surgical excision of the original primary
  * Mucosal melanoma
  * Stage IV melanoma (cutaneous, ocular, mucosal, or unknown primary)
* The following groups of patients may be entered onto this trial only if they are ineligible for S0008 or are, in the opinion of the managing physician, medically unfit to receive standard high-dose interferon:

  * Any clinically evident satellite or in-transit disease
  * Stage II disease with gross extracapsular extension
  * Recurrence in a previously resected nodal basin
  * Four or more involved lymph nodes or matted lymph nodes
  * Ulcerated primary melanoma and any involved lymph nodes

    * NOTE: Patients who are eligible for S0008 will be strongly encouraged to participate in that study in preference to this one
* Patients must have been surgically rendered free of disease with negative margins on resected specimens; patients rendered free of disease by non-surgical means are not eligible
* Patients must be randomized within 112 days (16 weeks) of surgical resection; if more than one surgical procedure is required to render the patient disease-free, all required surgeries must be accomplished within this 16 week time period
* Patients must not have received any adjuvant treatment (chemotherapy, biotherapy, or limb perfusion) after the resection(s) that make(s) them eligible for this trial; one systemic treatment after a prior surgery is allowed, and must have been completed >= 8 weeks prior to randomization; (when chemotherapy and biotherapy are given together as one planned treatment [biochemotherapy], this counts as one regimen); NOTE: Previous radiation therapy, including after the resection, is allowed as long as 30 days elapse between the radiation and initiation of therapy
* Prior treatment with GM-CSF or any peptides used in this protocol, is not allowed
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must not have an active infection requiring treatment with parenteral antibiotics
* Patients must not have other significant medical, surgical, or psychiatric conditions or require any medication or treatment that may interfere with compliance on any of the E4697 treatment regimens
* Patients must not have a diagnosis or evidence of organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the full protocol
* Patients must be able to self-administer or arrange for administration of subcutaneous injections
* Patients who have other current malignancies are not eligible
* Patients with prior history at any time of any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ are eligible; patients who meet this criteria must be disease-free at time of randomization
* Patients with prior history of basal or squamous skin cancer are eligible; patients who meet this criteria must be disease-free at time of randomization
* Patients who have had multiple primary melanomas are eligible
* Patients with other malignancies are eligible if they have been continuously disease free for > 5 years prior to the time of randomization
* Patients must not have autoimmune disorders, conditions of immunosuppression or treatment with systemic corticosteroids, including oral steroids (i.e., prednisone, dexamethasone), continuous use of topical steroid creams or ointments, or any steroid containing inhalers; replacement doses of steroids for patients with adrenal insufficiency are allowed; patients who discontinue use of these classes of medication for at least 2 weeks prior to randomization are eligible if, in the judgment of the treating physician, the patient is not likely to require these classes of drugs during the study
* Women of childbearing potential must not be pregnant (negative beta human chorionic gonadotropin [bHCG] within 2 weeks prior to randomization) or breast-feeding
* Women of childbearing potential and sexually active males must be counseled to use an accepted and effective method of contraception (including abstinence) while on treatment and for a period of 18 months after completing or discontinuing treatment
* All patients must have brain computed tomography (CT) or magnetic resonance imaging (MRI), chest CT or chest x-ray (CXR), and abdominal (liver) CT or MRI within 4 weeks prior to randomization; positron emission tomography (PET) scans are also acceptable in place of CT, CXR and/or abdominal MRI if obtained within 4 weeks prior to randomization; patients with lesions on the lower extremity must also have pelvic imaging within this time period; this is also strongly recommended for patients with lesions on the lower trunk; PET scans are acceptable
* Patients with resection of visceral disease must have imaging of the affected area/organ documenting disease-free status within 2 weeks prior to randomization
* White blood cells (WBC) >= 3,000/mm?
* Platelet count >= 100,000/mm?
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2 x institutional upper limit (IUL) of normal
* Bilirubin =< 2 x IUL of normal
* Serum creatinine =< 1.8 mg/dl
* Alkaline phosphatase and lactate dehydrogenase (LDH) must be performed within 4 weeks prior to randomization; LDH must be normal; patients with abnormal alkaline phosphatase which is =< 1.25 times the institutional upper limit of normal who have a negative CT or MRI of the liver and negative bone scan or a negative PET scan are eligible
* Patients with bone pain must have a bone scan within 4 weeks prior to randomization to document the absence of tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Actual)
Dates: Start 2000-02-23 (Actual); Primary Completion 2012-10-08 (Actual); Study Completion 2013-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Lawson, Principal Investigator — Eastern Cooperative Oncology Group
Locations (148):
- United States (148):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Veterans Administration-San Diego Medical Center, San Diego, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Southwest Florida Regional Medical Center, Fort Myers, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Florida Cancer Specialists-West Palm Beach, West Palm Beach, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Franklin Medical Center, Greenfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Saint John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - East Tennessee State University, Johnson City, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin

REFERENCES:
- [Derived] Lawson DH, Lee S, Zhao F, Tarhini AA, Margolin KA, Ernstoff MS, Atkins MB, Cohen GI, Whiteside TL, Butterfield LH, Kirkwood JM. Randomized, Placebo-Controlled, Phase III Trial of Yeast-Derived Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) Versus Peptide Vaccination Versus GM-CSF Plus Peptide Vaccination Versus Placebo in Patients With No Evidence of Disease After Complete Surgical Resection of Locally Advanced and/or Stage IV Melanoma: A Trial of the Eastern Cooperative Oncology Group-American College of Radiology Imaging Network Cancer Research Group (E4697). J Clin Oncol. 2015 Dec 1;33(34):4066-76. doi: 10.1200/JCO.2015.62.0500. Epub 2015 Sep 8. PMID 26351350
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open between December 29, 1999 and October 31, 2006. A total of 815 patients were enrolled.
Groups:
- Arm I (GM-CSF, Peptide Vaccine): Patients receive GM-CSF (sargramostim) SC on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  sargramostim: Given SC
  peptide vaccine: Given SC
- Arm II (GM-CSF Placebo, Peptide Vaccine): Patients receive GM-CSF (sargramostim) placebo SC on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  peptide vaccine: Given SC
  GM-CSF placebo: Given SC
- Arm III (GM-CSF, Peptide Placebo): Patients receive GM-CSF (sargramostim) SC on days 1-14 and peptide placebo mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  sargramostim: Given SC
  peptide placebo: Given SC
- Arm IV (GM-CSF Placebo, Peptide Placebo): Patients receive GM-CSF placebo SC on days 1-14 and peptide placebo on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  GM-CSF placebo: Given SC
  peptide placebo: Given SC
- Arm V (GM-CSF): Patients receive GM-CSF (sargramostim) SC on days 1-14.
  sargramostim: Given SC
- Arm VI (GM-CSF Placebo): Patients receive GM-CSF (sargramostim) placebo SC on days 1-14.
  GM-CSF placebo: Given SC
Period: Overall Study
Arm/Group | Arm I (GM-CSF, Peptide Vaccine) | Arm II (GM-CSF Placebo, Peptide Vaccine) | Arm III (GM-CSF, Peptide Placebo) | Arm IV (GM-CSF Placebo, Peptide Placebo) | Arm V (GM-CSF) | Arm VI (GM-CSF Placebo)
Started | 109 | 111 | 109 | 107 | 190 | 189
Treated | 104 | 110 | 107 | 104 | 186 | 171
Completed | 54 | 53 | 47 | 56 | 92 | 79
Not Completed | 55 | 58 | 62 | 51 | 98 | 110
Not completed — Lack of Efficacy | 35 | 48 | 48 | 43 | 71 | 79
Not completed — Adverse Event | 2 | 1 | 3 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 5 | 1 | 12 | 4
Not completed — complicating disease | 1 | 1 | 2 | 0 | 1 | 0
Not completed — error | 2 | 1 | 1 | 1 | 1 | 1
Not completed — maximum dose reached | 0 | 1 | 0 | 0 | 1 | 0
Not completed — unknown/not specify | 3 | 4 | 1 | 3 | 3 | 5
Not completed — not start protocol therapy | 5 | 1 | 2 | 3 | 4 | 18
Not completed — alternative therapy | 3 | 0 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All patients regardless of eligibility and treatment status
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (GM-CSF, Peptide Vaccine) | Arm II (GM-CSF Placebo, Peptide Vaccine) | Arm III (GM-CSF, Peptide Placebo) | Arm IV (GM-CSF Placebo, Peptide Placebo) | Arm V (GM-CSF) | Arm VI (GM-CSF Placebo) | Total
Number analyzed (Participants) | 109 | 111 | 109 | 107 | 190 | 189 | 815
Age, Continuous [Median (Full Range); unit: years] | 60 [27 to 83] | 56 [22 to 82] | 57 [23 to 87] | 58 [23 to 82] | 60 [19 to 88] | 57 [19 to 87] | 58 [19 to 88]
Sex/Gender, Customized [Number; unit: participants] — One patient on arm V had missing data for gender. Hence, a total of 189 patients on arm V reported gender.
  participants
    Female | 48 | 45 | 45 | 39 | 77 | 77 | 331
    Male | 61 | 66 | 64 | 68 | 112 | 112 | 483

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as time from randomization to death from any cause.
Time Frame: assessed every 3 months if patient is < 2 years from study entry and every 6 months if patient is 2-5 years from study entry, and annually if >5 years, up to year 15
Population: all randomized patients, regardless of eligibility
Measure: Median (95% Confidence Interval); unit: months
Groups:
- GM-CSF: Patients received GM-CSF in the trial, including patients on arms I, III, V.
- GM-CSF Placebo: Patients who did not receive GM-CSF (ie, received GM-CSF placebo) in the trial, including patients on arms II, IV and VI
Arm/Group | GM-CSF | GM-CSF Placebo
Number analyzed (Participants) | 408 | 407
months | 69.6 [53.4 to 83.5] | 59.3 [44.4 to 77.3]
Statistical Analysis 1: Comparison: GM-CSF vs GM-CSF Placebo; Test type: Superiority or Other; p = 0.528, Log Rank; stratifying on HLA-A2 status, site of metastases and number of metastatic lesions

2. Primary Outcome: Recurrence Free Survival
Description: Recurrence free survival is defined as time from randomization to first disease recurrence or death from any cause (whichever occur first), censoring cases without recurrence or death at the last date of known free of recurrence free survival events. Disease recurrence was determined based on positive cytology or biopsy in the presence of a single new lesion or the appearance of multiple lesions consistent with metastatic disease, or a positive brain CT or MRI scan or CSF cytology.
Time Frame: as for outcome 1
Population: all randomized patients, regardless of eligibility
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GM-CSF | GM-CSF Placebo
Number analyzed (Participants) | 408 | 407
months | 11.4 [9.4 to 14.8] | 8.8 [7.5 to 11.2]
Statistical Analysis 1: Comparison: GM-CSF vs GM-CSF Placebo; Test type: Superiority or Other; p = 0.131, Log Rank; stratifying on HLA-A2 status, site of metastases, and number of metastatic lesions

3. Secondary Outcome: Overall Survival in Human Leukocyte Antigens-A2 (HLA-A2) Positive Patients
Description: Overall survival is defined as time from randomization to death from any cause.
Time Frame: assessed every 3 months if patient is < 2 years from study entry and every 6 months if patient is 2-5 years from study entry, and annually if >5 years,up to year 15
Population: all HLA-A2 positive patients
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Peptide Vaccination: Patients who were HLA-A2 positive and received peptide vaccine in the trial, including 109 patients on arm I and 111 patients on arm II.
- Peptide Placebo: Patients who were HLA-A2 positive and received peptide placebo in the trial, including 109 patients on arms III and 107 patients on arm IV
Arm/Group | Peptide Vaccination | Peptide Placebo
Number analyzed (Participants) | 220 | 216
months | 68.6 [47.0 to 92.3] | 63.3 [49.2 to 105.0]
Statistical Analysis 1: Comparison: Peptide Vaccination vs Peptide Placebo; Test type: Superiority or Other; p = 0.60, Log Rank; stratifying on GM-CSF, site of metastases and number of metastatic lesions

4. Secondary Outcome: Recurrence Free Survival in HLA-A2 Positive Patients
Description: as for outcome 2
Time Frame: as for outcome 1
Population: all HLA-A2 positive patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Peptide Vaccination | Peptide Placebo
Number analyzed (Participants) | 220 | 216
months | 11.5 [8.7 to 20.4] | 9.8 [7.7 to 15.5]
Statistical Analysis 1: Comparison: Peptide Vaccination vs Peptide Placebo; Test type: Superiority or Other; p = 0.71, Log Rank — stratifying on GM-CSF, site of metastases and number of metastatic lesions

5. Secondary Outcome: 5-year Overall Survival Rate
Description: Overall survival is defined as time from randomization to death from any cause, and 5-year overall survival rate is estimated via Kaplan-Meier method.
Time Frame: as for outcome 1
Population: all randomized patients, regardless of eligibility
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (GM-CSF, Peptide Vaccine) | Arm II (GM-CSF Placebo, Peptide Vaccine) | Arm III (GM-CSF, Peptide Placebo) | Arm IV (GM-CSF Placebo, Peptide Placebo) | Arm V (GM-CSF) | Arm VI (GM-CSF Placebo)
Number analyzed (Participants) | 109 | 111 | 109 | 107 | 190 | 189
percentage of participants | 55.5 [45.4 to 64.5] | 51.9 [42.0 to 61.0] | 51.1 [41.2 to 60.1] | 51.6 [41.4 to 60.9] | 51.2 [43.8 to 58.2] | 46.7 [39.3 to 53.8]
Statistical Analysis 1: Comparison: Arm I (GM-CSF, Peptide Vaccine) vs Arm II (GM-CSF Placebo, Peptide Vaccine) vs Arm III (GM-CSF, Peptide Placebo) vs Arm IV (GM-CSF Placebo, Peptide Placebo); Treatment arm comparison in patients with positive HLA-A2 status; Test type: Superiority or Other; p = 0.88, Log Rank; stratifying on site of metastases and number of metastatic lesions
Statistical Analysis 2: Comparison: Arm V (GM-CSF) vs Arm VI (GM-CSF Placebo); Treatment arm comparison in patients with negative HLA-A2 status; Test type: Superiority or Other; p = 0.69, Log Rank; stratifying on site of metastases and number of metastatic lesions

6. Secondary Outcome: 5-year Recurrence Free Survival Rate
Description: Recurrence free survival is defined as time from randomization to first disease recurrence or death from any cause (whichever occur first), censoring cases without recurrence or death at the last date of known free of recurrence free survival events, and 5-year overall survival rate is estimated via Kaplan-Meier method. Disease recurrence was determined based on positive cytology or biopsy in the presence of a single new lesion or the appearance of multiple lesions consistent with metastatic disease, or a positive brain CT or MRI scan or CSF cytology.
Time Frame: as for outcome 1
Population: all randomized patients, regardless of eligibility
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (GM-CSF, Peptide Vaccine) | Arm II (GM-CSF Placebo, Peptide Vaccine) | Arm III (GM-CSF, Peptide Placebo) | Arm IV (GM-CSF Placebo, Peptide Placebo) | Arm V (GM-CSF) | Arm VI (GM-CSF Placebo)
Number analyzed (Participants) | 109 | 111 | 109 | 107 | 190 | 189
percentage of participants | 32.4 [23.6 to 41.5] | 33.2 [24.4 to 42.2] | 31.3 [22.8 to 40.2] | 28.0 [19.7 to 36.9] | 30.6 [24.1 to 37.3] | 22.9 [17.1 to 29.2]
Statistical Analysis 1: Comparison: Arm I (GM-CSF, Peptide Vaccine) vs Arm II (GM-CSF Placebo, Peptide Vaccine) vs Arm III (GM-CSF, Peptide Placebo) vs Arm IV (GM-CSF Placebo, Peptide Placebo); Treatment arm comparison in patients with positive HLA-A2 status; Test type: Superiority or Other; p = 0.91, Log Rank; stratifying on site of metastases and number of metastatic lesions
Statistical Analysis 2: Comparison: Arm V (GM-CSF) vs Arm VI (GM-CSF Placebo); Treatment arm comparisons in patients with negative HLA-A2 status; Test type: Superiority or Other; p = 0.13, Log Rank; stratifying on site of metastases and number of metastatic lesions

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 cycle=28 days) for cycles 1, 2, 3, and 4; after cycle 4, assessed every 3 months (at the completion of cycles 7, 10, 13) while on treatment and for 30 days after the end of treatment
Description: After off treatment, if the patient experienced any clinical problems possibly related to the protocol treatment, the clinical problems were also reported per the standard ECOG follow-up schedule: every 3 months if patient is <2 years from study entry, every 6 months if patient is 2-5 years from study entry, and every 12 months if >5 years.
Groups:
- Arm I (GM-CSF, Peptide Vaccine): Arm I (GM-CSF, peptide vaccine) Patients receive GM-CSF (sargramostim) SC on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  sargramostim: Given SC peptide vaccine: Given SC
- Arm II (GM-CSF Placebo, Peptide Vaccine): Arm II (GM-CSF placebo, peptide vaccine) Patients receive GM-CSF (sargramostim) placebo SC on days 1-14 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  peptide vaccine: Given SC GM-CSF placebo: Given SC
- Arm III (GM-CSF, Peptide Placebo): Arm III (GM-CSF, peptide placebo) Patients receive GM-CSF (sargramostim) SC on days 1-14 and peptide placebo mixed with either incomplete Freund's adjuvant or Montanide ISA-51 VG SC on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  sargramostim: Given SC peptide placebo: Given SC
- Arm IV (GM-CSF Placebo, Peptide Placebo): Arm IV (GM-CSF placebo, peptide placebo) Patients receive GM-CSF placebo SC on days 1-14 and peptide placebo on days 1 and 15 (course 1) and day 1 (course 2 and subsequent courses).
  GM-CSF placebo: Given SC peptide placebo: Given SC
Arm/Group | Arm I (GM-CSF, Peptide Vaccine) | Arm II (GM-CSF Placebo, Peptide Vaccine) | Arm III (GM-CSF, Peptide Placebo) | Arm IV (GM-CSF Placebo, Peptide Placebo) | Arm V (GM-CSF) | Arm VI (GM-CSF Placebo)
Serious Adverse Events (participants affected / at risk) | 12/104 | 17/110 | 15/107 | 9/104 | 22/186 | 12/171
Other Adverse Events (participants affected / at risk) | 104/104 | 109/110 | 105/107 | 102/104 | 180/186 | 143/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (GM-CSF, Peptide Vaccine) (N=104) | Arm II (GM-CSF Placebo, Peptide Vaccine) (N=110) | Arm III (GM-CSF, Peptide Placebo) (N=107) | Arm IV (GM-CSF Placebo, Peptide Placebo) (N=104) | Arm V (GM-CSF) (N=186) | Arm VI (GM-CSF Placebo) (N=171)
Anaphylaxis (Immune system disorders) | 1 | 1 | 1 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
White blood cell decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 2 | 2 | 2 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 3 | 0 | 1 | 1
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 2 | 9 | 2 | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 3 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, spe (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — infection with grade 3 or 4 neutropenia
Infections and infestations - Other, spe (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 — infection with unknown ANC
Infections and infestations - Other, spe (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — infection w/o neutropenia
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue di (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, specif (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 1 | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
Flushing (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (GM-CSF, Peptide Vaccine) (N=104) | Arm II (GM-CSF Placebo, Peptide Vaccine) (N=110) | Arm III (GM-CSF, Peptide Placebo) (N=107) | Arm IV (GM-CSF Placebo, Peptide Placebo) (N=104) | Arm V (GM-CSF) (N=186) | Arm VI (GM-CSF Placebo) (N=171)
Anemia (Blood and lymphatic system disorders) | 21 | 15 | 26 | 18 | 25 | 16
White blood cell decreased (Investigations) | 7 | 9 | 8 | 12 | 7 | 13
Neutrophil count decreased (Investigations) | 3 | 10 | 5 | 10 | 8 | 11
Platelet count decreased (Investigations) | 6 | 4 | 8 | 2 | 5 | 6
Cardiac disorders - Other, specify (Cardiac disorders) | 6 | 4 | 9 | 7 | 6 | 5
Fatigue (General disorders) | 67 | 53 | 58 | 57 | 81 | 66
Fever (General disorders) | 17 | 19 | 15 | 6 | 21 | 13
Chills (General disorders) | 24 | 13 | 14 | 7 | 24 | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 4 | 4 | 6 | 11 | 7
Weight gain (Investigations) | 7 | 6 | 6 | 10 | 7 | 8
Weight loss (Investigations) | 2 | 7 | 5 | 6 | 8 | 8
General disorders and administration sit (General disorders) | 5 | 6 | 6 | 5 | 8 | 5
Bruising (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 6 | 3 | 4
Injection site reaction (General disorders) | 99 | 100 | 98 | 89 | 147 | 43
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 10 | 15 | 5 | 17 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27 | 22 | 33 | 13 | 31 | 17
Skin and subcutaneous tissue disorders - (Skin and subcutaneous tissue disorders) | 15 | 16 | 11 | 14 | 22 | 6
Hot flashes (Vascular disorders) | 3 | 1 | 6 | 3 | 10 | 3
Anorexia (Metabolism and nutrition disorders) | 7 | 7 | 6 | 7 | 17 | 9
Nausea (Gastrointestinal disorders) | 24 | 24 | 21 | 15 | 36 | 19
Dysgeusia (Nervous system disorders) | 3 | 2 | 5 | 4 | 10 | 4
Vomiting (Gastrointestinal disorders) | 6 | 5 | 5 | 4 | 8 | 3
Diarrhea (Gastrointestinal disorders) | 16 | 8 | 11 | 11 | 27 | 19
Alkaline phosphatase increased (Investigations) | 7 | 5 | 3 | 10 | 9 | 15
Blood bilirubin increased (Investigations) | 5 | 4 | 9 | 3 | 9 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 | 14 | 20 | 15 | 24 | 18
Aspartate aminotransferase increased (Investigations) | 5 | 7 | 2 | 7 | 14 | 12
Dizziness (Nervous system disorders) | 5 | 1 | 4 | 6 | 7 | 8
Insomnia (Psychiatric disorders) | 3 | 2 | 5 | 6 | 9 | 9
Anxiety (Psychiatric disorders) | 2 | 4 | 6 | 5 | 8 | 2
Depression (Psychiatric disorders) | 3 | 3 | 2 | 6 | 10 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4 | 6 | 13 | 10 | 7
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 3 | 3 | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 23 | 32 | 18 | 37 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 11 | 14 | 7 | 15 | 10
Non-cardiac chest pain (General disorders) | 0 | 1 | 3 | 0 | 10 | 1
Headache (Nervous system disorders) | 28 | 24 | 22 | 21 | 42 | 36
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 32 | 38 | 25 | 57 | 26
Pain (General disorders) | 8 | 9 | 5 | 10 | 10 | 11
Creatinine increased (Investigations) | 5 | 6 | 5 | 8 | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less